CLINICAL TRIAL: NCT00064324
Title: A Phase II Study of Perifosine in Soft Tissue Sarcoma
Brief Title: Perifosine in Treating Patients With Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02798; MC0276; 5972; N01CM17104 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Adult Soft Tissue Sarcoma; Stage III Adult Soft Tissue Sarcoma; Stage IV Adult Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — perifosine; octadecyl-(N,N-dimethylpiperidino-4-yl)-phosphate

ARMS (1):
- Arm I (Experimental): Patients receive a loading dose of oral perifosine every 6 hours for a total of 4 doses on day 1 and once daily on days 2-28 of course 1 only. For all subsequent courses, patients receive oral perifosine once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: perifosine; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: perifosine — Given orally
  Other Names: D21266; octadecylphosphopiperidine
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase II trial to study the effectiveness of perifosine in treating patients who have advanced soft tissue sarcoma. Drugs used in chemotherapy such as perifosine use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the 6-month progression-free rate in patients treated with perifosine and having advanced soft tissue sarcoma.

SECONDARY OBJECTIVES:

I. To evaluate survival and time to progression. II. To evaluate objective tumor response status and duration. III. To evaluate adverse event rates. IV. To evaluate patterns of treatment failure. V. To evaluate pharmacokinetics.

OUTLINE: This is a multicenter study.

Patients receive a loading dose of oral perifosine every 6 hours for a total of 4 doses on day 1 and once daily on days 2-28 of course 1 only. For all subsequent courses, patients receive oral perifosine once daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 5 years.

PROJECTED ACCRUAL: A total of 17-46 patients will be accrued for this study within 9-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced soft tissue sarcoma
* Measurable disease; measurable disease lesions that are being monitored for response and have been previously irradiated must have progressed > 25% since completion of radiation therapy
* Absolute neutrophil count (ANC) >= 1,500/uL
* PLT >= 100,000/uL
* Total bilirubin =< upper normal limit (UNL)
* AST =< 2.5 x UNL
* Creatinine =< UNL or calculated creatinine clearance >= 60 mL/min (i.e. using the Cockcroft-Gault or Jeliffe methods)
* Life expectancy >= 12 weeks
* ECOG performance status (PS) 0 or 1
* Capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent

Exclusion Criteria:

* Any of the following as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Breastfeeding women
  * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
  * NOTE: Pregnant women are excluded from this study because perifosine is an alkylphospholipid with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with perifosine, breastfeeding should be discontinued if the mother is treated with perifosine
* Any of the following:

  * >= 3 prior cytotoxic chemotherapy regimens for metastatic sarcoma
  * Chemotherapy =< 4 weeks prior to study entry
  * Nitrosoureas or mitomycin C =< 6 weeks prior to study entry
  * Radiotherapy =< 4 weeks prior to study entry
  * Immunotherapy =< 4 weeks prior to study entry
  * Biologic therapy =< 4 weeks prior to study entry
  * Failure to recover from acute, reversible effects of prior therapy regardless of interval since last treatment
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-FDA-approved indication and in the context of a research investigation)
* Uncontrolled brain metastases; NOTE: these patients are excluded because of the poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; however, if brain metastasis are treated and controlled for > 8 weeks, the patient would be eligible for this study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic cardiac arrhythmia despite appropriate therapy, or psychiatric illness/social situations that would limit compliance with study requirements
* HIV-positive patients receiving combination anti-retroviral therapy; NOTE: these patients are excluded from the study because of possible pharmacokinetic interactions with perifosine; appropriate studies may be undertaken in patients receiving combination anti-retroviral therapy when indicated
* Prior malignancy, except for the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * Adequately treated noninvasive carcinoma
  * Other invasive cancer from which the patient has been disease-free for 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2003-06; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Progression-free rate | 6 months

SECONDARY OUTCOMES:
Survival time | Time from regstration to death due to any cause, assessed up to 5 years
  Estimated using the method of Kaplan-Meier (Kaplan and Meier 1958) and Cox Proportional Hazards (Cox D. 1972) modeling.
Time to disease progression | Time from registration to documentation of disease progression, assessed up to 5 years
  Estimated using the method of Kaplan-Meier (Kaplan and Meier 1958) and Cox Proportional Hazards (Cox D. 1972) modeling.
Duration of response | Date at which the patient's objective status is first noted to be either a complete response (CR) or partial response (PR) to the date progression is documented, assessed up to 5 years
Time to treatment failure | Time from the date of randomization to the date at which the patient is removed from treatment due to progression, toxicity, or refusal, assessed up to 5 years
Average change over time for PK variable(s) | Days 1 and 15 of course 1 and day 1 of courses 2-6
  Estimated and tested via appropriate methods (i.e. t-test or Wilcoxon tests).

CONTACTS AND LOCATIONS:
Overall Officials: Howard Bailey, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States